CLINICAL TRIAL: NCT04794075
Title: Programme d'Éducation Thérapeutique et d'Accompagnement Infirmier Vers Les Soins de Support, Chez Les Patientes Sous Hormonothérapie Pour un Cancer du Sein Non métastatique
Brief Title: Therapeutic Education and Nursing Support Program for Supportive Care, in Patients Treated With Hormone Therapy for Non-metastatic Breast Cancer
Acronym: ETAPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other); Walisco (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH2_BREYSSE_ETAPH; 2020-A03074-35 (Registry Identifier: IRCB)
Record Dates: First submitted 2021-02-22; First posted 2021-03-11 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Neoplasm of Breast
Keywords: Therapeutic Education; Nursing Support Program; Hormone Therapy; Non-metastatic Breast Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Quasi-experiment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group with the therapeutic education and nursing support program (Experimental): In addition to the conventional oncology follow-up, patients will participate in an initial educational assessments day.
  Interventions: Other: Therapeutic Education and Nursing Support Program for Supportive Care
- Control group (No Intervention): Patients will have the conventional oncology follow-up.

INTERVENTIONS:
Other: Therapeutic Education and Nursing Support Program for Supportive Care — In addition to the conventional oncology follow-up, patients will participate in an initial educational assessment day within 15 days before or after their first dose of hormone therapy.
  A discussion between the patient and the pivot nurse will then make it possible to define personalized objectives, thus guiding the choice of workshops in the outpatient educational program.
  Arms: Experimental group with the therapeutic education and nursing support program

SUMMARY:
To compare the efficacy of the addition of a therapeutic education program combined with nursing phone follow-up, compared to conventional management alone, on the management of adverse events (AEs) related to adjuvant hormone therapy during the first year of treatment in patients with non-metastatic breast cancer.

DETAILED DESCRIPTION:
The main objective of the ETAPH project is to offer breast cancer patients multidisciplinary care that will limit the impact of adverse effects related to hormone therapy treatment and improve their quality of life. The achievement of this objective is based on therapeutic education and nursing follow-up throughout the first year of treatment, which, thanks to active listening and coordination of the various players, will enable global and personalized patient care.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 75 years inclusive
* Patients with non-metastatic breast cancer for whom adjuvant hormone therapy (anti-oestrogen or anti-aromatase) is indicated, depending on the decision of the multidisciplinary consultation meeting.
* Performance status (ECOG) ≤ 2
* Patient able to read and understand French (common use)
* Patient with access to an internet connection (for collection of adverse events and responses to questionnaires on the electronic platform)
* Patient who has been informed and has given written consent to participate in the study
* Patient affiliated to the French social security system or equivalent

Exclusion Criteria:

* Patient with metastatic cancer (stage IV)
* Patient undergoing neoadjuvant hormone therapy
* Patient who started hormone therapy prior to inclusion in the study
* Patient with a history of other cancer treated by radiotherapy, chemotherapy or hormone therapy, with an end of treatment less than 2 years ago.
* For patients in the experimental group: Inability of the patient to travel to the hospital to attend the initial assessment day and the proposed group outpatient workshops; follow-up of the program difficult for geographical, physical or other reasons (at the discretion of the investigator).
* For patients in the control group: patients for whom telephone nursing follow-up is planned for 2 months or more or more than 4 sessions of therapeutic education.
* Pregnant and breastfeeding women
* Patient with a documented history of cognitive or psychiatric disorders
* Refusal to participate, protected adult patient, under guardianship or curatorship

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of adding a therapeutic education program combined with nursing phone follow-up, compared to conventional management alone on the management of adverse events related to adjuvant hormone therapy. | For a year
  The primary endpoint is the score of the 7 adverse events (AEs), graded on a Likert scale from 0 to 4 points from the NCI-CTCAE v5.0, which will be transformed into a single composite endpoint.
  The 7 AEs considered here will be the most frequent and troublesome of the hormone therapy, namely: muscle and/or joint pain, hot flashes, headache, fatigue, insomnia/sleep disturbance, weight gain, nausea. This collection will be done initially (T0) and then monthly by the patients.

SECONDARY OUTCOMES:
To compare the effectiveness of adding the program to conventional management alone in terms of quality of life for patients on hormone therapy at baseline (Day 0), Month 6 and Month 12. | Change from baseline at Month 6 and Month 12
  The score of the validated Quality of Life of Cancer Patients (EORTC-QLQ-C30) self-questionnaire score, performed at Day 0, Month 6 and Month 12 after initiation of hormone therapy
To compare the effectiveness of adding the program to conventional management alone in terms of sleep quality at baseline (Day 0), Month 6 and Month 12. | Change from baseline at Month 6 and Month 12
  the score of the validated Pittsburgh sleep quality self-questionnaire during the past month, performed at Day 0, Month 6 and Month 12 after initiation of hormone therapy
To compare the effectiveness of adding the program to conventional management alone in terms of drug use for the management of adverse events throughout the study. | From date of first Hormone Therapy intake to 12 months
  The INN name,the daily dosage and duration (number of days) of medication taken between Day 0 and 12 months, will be assessed to compare between the experimental ans the control group in term of medication use
To compare the effectiveness of adding the program to conventional management alone in terms of therapeutic compliance at Month 6 and Month 12. | Change from Month 6 and Month 12
  GIRERD's subjective compliance self-questionnaire score will be filled in at Month 6 and Month 12.
To compare the effectiveness of adding the program to conventional management alone in terms of patients' confidence regarding the use of hormone therapy at Day 0, Month 6 and Month 12. | Change from baseline at Month 6 and Month 12
  Patients' confidence in their treatment, assessed on a numerical scale from 0 to 10, measured at Day 0, Month 6 and Month 12.
To compare the effectiveness of adding the program to conventional management alone in terms of patients' level of knowledge about the disease and treatment. | Change from baseline at Month 2
  Score obtained in the knowledge quizz conducted in Day 0, then at 2 months. This questionnaire is developed by our team based on Likert scales from 1 to 4.
To compare the effectiveness of adding the program to conventional management alone in terms of patients' satisfaction with their care at Month 12. | For a year
  Score of satisfaction with patient care in relation to the needs they have had over the past 12 months. This questionnaire is developed by our team based on Likert scales from 0 to 3.
To compare the effectiveness of adding the program to conventional management alone in terms of medico-economic impact of the program, in terms of cost-utility. | For a year
  the cost-utility ratio of the program will be calculated by estimating the costs incurred/avoided by this program and the evolution of the quality of life of the patients at different times.
To assess patient interest in and adherence to the proposed program in the experimental group. | For a year
  Refusal rate and program participation rate The rate of premature exit or loss of sight The number and type of workshops attended by patients Evaluation of program content based on Likert scales ranging from 1 to 4.
To describe the non-drug means used by patients to manage their adverse events and their use of supportive care during the study. | For a year
  Patients' non-drug management of side effects and use of supportive care will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Breysse, Principal Investigator — Centre Hospitalier Emile Roux
Locations (9):
- France (9):
  - Centre Hospitalier de Bourg-en-Bresse / Fleyriat, Bourg-en-Bresse
  - Clinique De L'infirmerie Protestante De Lyon, Caluire-et-Cuire
  - CH de Carcassonne, Carcassonne
  - CHAL - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Centre Hospitalier François Quesnay, Mantes-la-Jolie
  - Groupement Hospitalier Portes de Provence, Montélimar
  - Centre Hospitalier Universitaire de Saint-Étienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Médipôle Lyon-Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No
The study sponsor is the owner of the data and no use or transmission to a third party may be made without its prior consent. All information resulting from this clinical research protocol is considered confidential.